CLINICAL TRIAL: NCT06116617
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SRSD107 in Healthy Participants
Brief Title: A Phase 1 Study to Evaluate the Safety, Tolerability, PK/PD of SRSD107 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirius Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SRSD107-101
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRSD107 (Experimental): SRSD107 for subcutaneous (s.c.) injection Group A1, 15mg, single dose Group A2, 45mg, single dose Group A3, 120mg, single dose Group A4, 240mg, single dose Group A5, 450mg, single dose
  Interventions: Drug: SRSD107
- Placebo (Placebo Comparator): Sodium chloride for subcutaneous (s.c.) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRSD107 — SRSD107 is a synthetic, chemically modified double-stranded, small interfering ribonucleic acid (siRNA).
  Arms: SRSD107
Drug: Placebo — Sodium chloride
  Arms: Placebo

SUMMARY:
The primary aim of this study is to evaluate safety and tolerability data when SRSD107 is administered as single SC injections to healthy participants. This information, along with PK/PD data, will help establish the appropriate doses and dosing regimen for future studies in patients.

DETAILED DESCRIPTION:
SRSD107 is a synthetic, chemically modified double-stranded, small interfering ribonucleic acid (siRNA). The antisense strand is specifically designed to recognize and cleave human factor XI (FXI) messenger ribonucleic acid (mRNA) which reduces FXI protein. FXI protein reduction may prevent thromboembolic events without increasing the risk of bleeding.

This study will be a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study conducted in two parts. A total of 40 participants will be studied in 5 groups (Groups A1 to A5), each group consisting of 8 participants. In each group, 6 participants will receive SRSD107 and 2 will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, based on no clinically significant findings from medical history, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations.
* Activated partial thromboplastin time and PT within the normal range.
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
* Able to understand and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History or evidence of any abnormal bleeding or coagulation disorder; or evidence of coagulopathy, prolonged or unexplained, clinically significant bleeding, or frequent unexplained bruising or thrombus formation; or a history of spontaneous bleeding.
* Evidence of an active or suspected cancer, or a history of malignancy, within 5 years prior to screening. Nonmelanoma skin cancer, curatively treated localized prostate cancer, or other carcinoma in situ are not exclusionary, providing that they did not require systemic therapy and are considered cured.
* Acute of febrile illness within 7 days prior to dose administration or evidence of active infection.
* Any major surgery within 3 months prior to screening or plan to have any surgery during the study.
* History of clinically significant hypersensitivity, intolerance, or allergy to any drug compound, oligonucleotide, GalNAc, food, or other substance, as determined by the investigator (or designee).
* Confirmed systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg.
* QT interval corrected for heart rate using Fridericia's method (QTcF) >450 ms in males or >470 ms in females confirmed by repeat measurement.
* White blood cell count <3.5 × 109/L, platelets <100 × 109/L, or hemoglobin below the lower limit of normal.
* Alanine aminotransferase, aspartate aminotransferase, gamma glutamyl transferase, alkaline phosphatase, or total bilirubin >1.5 × the upper limit of normal (ULN).
* Estimated glomerular filtration rate <80 mL/min/1.73m2, as calculated by the 2021 Chronic Kidney Disease Epidemiology Collaboration equation.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Positive pregnancy test at screening or check in.
* Receipt of blood products within 2 months prior to check in.
* Loss of >500 mL whole blood or donation of blood products within 1 month prior to screening.
* History of intolerance to SC injections, or scarring (eg, from surgical procedures or burns) in areas when SC dose administration may occur.
* Participants who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of adverse events (AEs) | up to 168 days post last dose
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Proportion of Serious Adverse Events (SAEs) | up to 168 days post last dose
  A serious AE (SAE) is defined as any untoward medical occurrence that at any dose either:
  * results in death
  * is life threatening
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity (disability is defined as a substantial disruption of a person's ability to conduct normal life functions)
  * results in a congenital anomaly/birth defect
  * results in an important medical event (see below).

SECONDARY OUTCOMES:
Cmax | Group A, Day 1 to Day 3; Group B, Day 1 to Day 3 and Day 29 to 31
  Maximum observed plasma concentration
tmax | Group A, Day 1 to Day 3; Group B, Day 1 to Day 3 and Day 29 to 31
  Time to maximum plasma concentration
t1/2 | Group A, Day 1 to Day 3; Group B, Day 1 to Day 3 and Day 29 to 31
  Plasma half-life
AUC | Group A, Day 1 to Day 3; Group B, Day 1 to Day 3 and Day 29 to 31
  Area under the plasma concentration-time curve from 0 to infinity
CL/F | Group A, Day 1 to Day 3; Group B, Day 1 to Day 3 and Day 29 to 31
  Apparent total clearance
Effect of SRSD107 on circulating FXI Levels | up to 168 days post last dose
  Determination of % Lowering of FXI to Baseline FXI Level
Effect of SRSD107 on coagulation | up to 168 days post last dose
  Determination of % APTT to baseline APTT

CONTACTS AND LOCATIONS:
Overall Officials: Qiuyue Qu, Study Director — Sirius Therapeutics Co., Ltd.
Locations (1):
- Linear Clinical Research, Perth, Other (Non U.s.), Australia

IPD SHARING:
Plan to Share IPD: No